CLINICAL TRIAL: NCT04196335
Title: I Can sEe Left Atrial Appendage (ICELAA) Clinical Study
Acronym: ICELAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2459
Record Dates: First submitted 2019-11-05; First posted 2019-12-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2022-06

CONDITIONS: Efficacy, Self; Safety Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm (Experimental)
  Interventions: Device: intra-procedural intracardiac echocardiography

INTERVENTIONS:
Device: intra-procedural intracardiac echocardiography — use of intra-procedural intracardiac echocardiography during Watchman FLX devices
  Other Names: Watchman FLX Device

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of using intra-procedural intracardiac echocardiography (ICE) for WATCHMAN FLX Device implants in subjects with non-valvular atrial fibrillation to reduce the risk of stroke.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is of legal age to participate in the study per the laws of their respective geography;
2. The subject has documented paroxysmal, persistent, permanent or long-term/longstanding persistent non-valvular atrial fibrillation (i.e., the subject does not have mitral stenosis or a mechanical heart valve);the subject has not been diagnosed with rheumatic mitral valvular heart disease);
3. The subject is deemed by the treating physician to be suitable for the protocol defined pharmacologic regimens;
4. The subject has a calculated CHA2DS2-VASc score of 2 or greater;
5. The subject is able to undergo ICE examinations;The subject is able to undergo ICE(which will be used during the index procedure) and TEE (which will be performed at 45 days and may also be performed at baseline);
6. The subject is able to understand and willing to provide written informed consent to participate in the trial;
7. The subject is able and willing to return for required follow-up visits and examinations.

Exclusion Criteria:

1. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance must be brought to the attention of the sponsor to determine eligibility, regardless of type of co-enrollment being proposed;
2. The subject requires long-term anticoagulation therapy for reasons other than AF-related stroke risk reduction, for example due to an underlying hypercoaguable state (i.e., even if the device is implanted, the subjects would not be eligible to discontinue OAC due to other medical conditions requiring chronic warfarin therapy);
3. The subject has a history of atrial septal repair or has an ASD/PFO device;
4. The subject has an implanted mechanical valve prosthesis in any position;
5. The subject currently or has had any documented history of, New York Heart Association Class IV Congestive Heart Failure;
6. The subject is of childbearing potential and is or plans to become pregnant during the time of the study (method of assessment upon study physician's discretion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Rate of Device Leak | 45 days
  Rate of significant leak (>5 mm) as assessed by TEE at 45 days' post-implant.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Erik Nielsen-Kudsk, MD, Principal Investigator — Aarhus University Hospital Skejby
Locations (7):
- Aarhus Universitetshospital, Skejby, Denmark
- Italy (4):
  - Fondazione Toscana Gabriele Monasterio, Massa
  - Ospedale dell'Angelo, Mestre
  - Centro Cardiologico Fondazione Monzino, Milan
  - Ospedale San Bortolo, Vicenza
- Hospital de Sant Pau, Barcelona, Spain
- John Radcliffe, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen-Kudsk JE, Berti S, Caprioglio F, Ronco F, Arzamendi D, Betts T, Tondo C, Christen T, Allocco DJ. Intracardiac Echocardiography to Guide Watchman FLX Implantation: The ICE LAA Study. JACC Cardiovasc Interv. 2023 Mar 27;16(6):643-651. doi: 10.1016/j.jcin.2022.10.024. Epub 2023 Feb 8. PMID 36764917